CLINICAL TRIAL: NCT03024450
Title: Efficacy and Prognostic Factors of Trastuzumab Based Therapy in HER2 Positive Advanced Gastric Cancer: a Single Center Prospective Observational Study
Brief Title: Trastuzumab Based Therapy in HER2 Positive AGC
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tianshu Liu, Chief doctor and director of Department of medical oncology, Shanghai Zhongshan Hospital
Other Study IDs: ZS-ON-08
Record Dates: First submitted 2017-01-02; First posted 2017-01-18 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Gastric Adenocarcinoma
Keywords: Gastric cancer; HER2; trastuzumab; prognosis
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Biospecimen Retention: Samples Without DNA — spicimen with paraffin-embedded obtained by gastroscope or surgery
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HER2 positive AGC treated with H+CT: HER2 expression was assessed by IHC first. In the cases with IHC 2+, fluorescence in situ hybridization (FISH) was used to detect HER2/neu amplification levels. Only patients with high level of HER2 expression (IHC 3+ or IHC 2+ plus FISH positive) were eligible in this study.
  Interventions: Drug: H+CT

INTERVENTIONS:
Drug: H+CT — All patients were treated with trastuzumab plus chemotherapy as the first-line therapy. There were no protocol-specified chemotherapy regimens. This is a prospective observational study. Efficacy and safety of trastuzumab were analyzed, clinical and pathological data were collected to evaluate the potential prognostic factors on progressive free survival.
  Other Names: trastuzumab plus chemotherapy

SUMMARY:
Trastuzumab plus chemotherapy is an effective therapy in HER2 positive advanced gastric cancer (AGC). However, the efficacy of routine trastuzumab therapy and its association with clinicopathologic factors remain unclear. The object of the study is to determine whether the addition of trastuzumab to first-line chemotherapy improves efficacy compared with chemotherapy alone in HER2 positive AGC.

DETAILED DESCRIPTION:
A total of 98 patients with HER2 positive AGC were enrolled in this prospective observational study. All patients were treated with trastuzumab plus chemotherapy as the first line therapy. Efficacy and safety of trastuzumab were analyzed, clinical and pathological data were collected to evaluate the potential prognostic factors on progressive free survival.

ELIGIBILITY:
Inclusion Criteria:

1. pathology and medical imageology proven advanced gastric adenocarcinoma, inoperable;
2. received trastuzumab plus chemotherapy as the first-line palliative chemotherapy;
3. with measurable lesion with a diameter 20 mm using conventional computed tomography (CT) or magnetic resonance imaging (MRI) scans or 10 mm using spiral CT scans;
4. Eastern Cooperative Oncology Group performance status (ECOG PS ) of 0-2;
5. left ventricular ejection fraction(LVEF) more than 50 percents;
6. sufficient bone marrow, liver and renal function.

Exclusion Criteria:

1. received previous systemic therapy for advanced disease (except adjuvant/neoadjuvant chemotherapy completed at least 6 months before enrollment);
2. trastuzumab based adjuvant/neoadjuvant therapy;
3. treatment with any other anticancer therapy (lapatinib, immunotherapy, etc);
4. patients with heart failure, coronary artery disease or myocardial infarction within the previous 6 months.
5. trastuzumab based first line therapy started beyond 4 weeks from the first diagnoses of AGC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with HER2 positive advanced or metastatic gastric adenocarcinoma in Shanghai Zhongshan Hospital, Fu Dan University were prospectively collected. HER2 expression was assessed by IHC first. In the cases with IHC 2+, fluorescence in situ hybridization (FISH) was used to detect HER2/neu amplification levels.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2012-01; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
OS | 8 years
  OS was defined as time from the beginning of first line therapy to death
PFS | 8 years
  PFS was measured from the start of first line therapy to the date of progressive disease or death, with censoring of patients who were lost to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu / Liu, Doctor, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210
- [Result] Halon A, Donizy P, Biecek P, Rudno-Rudzinska J, Kielan W, Matkowski R. HER-2 expression in immunohistochemistry has no prognostic significance in gastric cancer patients. ScientificWorldJournal. 2012;2012:941259. doi: 10.1100/2012/941259. Epub 2012 May 3. PMID 22645475
- [Result] Shitara K, Yatabe Y, Matsuo K, Sugano M, Kondo C, Takahari D, Ura T, Tajika M, Ito S, Muro K. Prognosis of patients with advanced gastric cancer by HER2 status and trastuzumab treatment. Gastric Cancer. 2013 Apr;16(2):261-7. doi: 10.1007/s10120-012-0179-9. Epub 2012 Jul 14. PMID 22797858
- [Result] Gomez-Martin C, Lopez-Rios F, Aparicio J, Barriuso J, Garcia-Carbonero R, Pazo R, Rivera F, Salgado M, Salud A, Vazquez-Sequeiros E, Lordick F. A critical review of HER2-positive gastric cancer evaluation and treatment: from trastuzumab, and beyond. Cancer Lett. 2014 Aug 28;351(1):30-40. doi: 10.1016/j.canlet.2014.05.019. Epub 2014 Jun 3. PMID 24943493
- [Result] Gong J, Liu T, Fan Q, Bai L, Bi F, Qin S, Wang J, Xu N, Cheng Y, Bai Y, Liu W, Wang L, Shen L. Optimal regimen of trastuzumab in combination with oxaliplatin/ capecitabine in first-line treatment of HER2-positive advanced gastric cancer (CGOG1001): a multicenter, phase II trial. BMC Cancer. 2016 Feb 8;16:68. doi: 10.1186/s12885-016-2092-9. PMID 26857702
- [Result] Jiang H, Li Q, Yu S, Yu Y, Wang Y, Li W, Cui Y, Liu T. Impact of HER2 expression on outcome in gastric cancer patients with liver metastasis. Clin Transl Oncol. 2017 Feb;19(2):197-203. doi: 10.1007/s12094-016-1523-z. Epub 2016 Jun 20. PMID 27324991
- [Result] Aizawa M, Nagatsuma AK, Kitada K, Kuwata T, Fujii S, Kinoshita T, Ochiai A. Evaluation of HER2-based biology in 1,006 cases of gastric cancer in a Japanese population. Gastric Cancer. 2014 Jan;17(1):34-42. doi: 10.1007/s10120-013-0239-9. Epub 2013 Feb 22. PMID 23430266
- [Derived] Li Q, Li H, Jiang H, Feng Y, Cui Y, Wang Y, Ji Y, Yu Y, Li W, Xu C, Yu S, Zhuang R, Liu T. Predictive factors of trastuzumab-based chemotherapy in HER2 positive advanced gastric cancer: a single-center prospective observational study. Clin Transl Oncol. 2018 Jun;20(6):695-702. doi: 10.1007/s12094-017-1772-5. Epub 2017 Nov 22. PMID 29168107